CLINICAL TRIAL: NCT07271511
Title: Comparative Analysis of Postoperative Pain Following Single vs Multiple-Visit Root Canal Therapy in Single-Rooted Teeth of Diabetic Patients: A Randomized Controlled Trial
Brief Title: Postoperative Pain After Single vs Multiple-Visit Root Canal Treatment in Diabetic Patients
Acronym: RCT-DM-Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Faiz ur rahman, Postgraduate Resident, Department of Operative Dentistry, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCD-Endo-DM-001
Record Dates: First submitted 2025-11-22; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus; Postoperative Pain After Endodontic Treatment
Keywords: Single-Visit Endodontics; Multiple-Visit Endodontic; Root canal therapy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group randomized controlled trial. Participants are assigned to receive either the single-visit or multiple-visit root canal therapy and are followed identically over the same time period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Visit RCT (Experimental): Participants in this arm receive the complete root canal therapy procedure in a single clinical appointment. This includes local anesthesia, rubber dam isolation, access cavity preparation, biomechanical cleaning and shaping of the root canal system, and final obturation (filling) of the canal
  Interventions: Procedure: Single-Visit Root Canal Therapy
- Multiple-Visit RCT (Active Comparator): Participants in this arm receive root canal therapy over two separate appointments. The first visit includes local anesthesia, rubber dam isolation, access cavity preparation, and biomechanical cleaning and shaping of the root canal system, followed by the placement of an intracanal medication and a temporary restoration. The second visit involves the removal of the temporary material and the final obturation (filling) of the canal
  Interventions: Procedure: Single-Visit Root Canal Therapy; Procedure: Multiple-Visit Root Canal Therapy

INTERVENTIONS:
Procedure: Single-Visit Root Canal Therapy — A standard non-surgical root canal treatment protocol where the entire procedure-from access opening and canal instrumentation to final obturation-is completed in one continuous session, without the use of inter-appointment intracanal medication
Procedure: Multiple-Visit Root Canal Therapy — A standard non-surgical root canal treatment protocol performed over two clinical appointments. The first visit involves canal preparation and dressing with an intracanal medicament. The final visit, scheduled after an interim period, involves the removal of the medicament and the completion of the root canal filling.
  Arms: Multiple-Visit RCT

SUMMARY:
A short description of the clinical study, including a brief statement of the clinical study's hypothesis, written in language intended for the lay public.

DETAILED DESCRIPTION:
This study compares post-treatment pain after root canal therapy done in one visit versus two visits for patients with diabetes. Root canal treatment can sometimes cause pain afterwards, and it is unclear if the number of visits makes a difference, especially for diabetic patients who may have different healing and pain responses. We will randomly assign 200 diabetic patients needing a root canal on a single-rooted tooth to either have the entire procedure completed in a single appointment or split over two appointments. Patients will record their pain levels on a standard scale at 24 hours, 72 hours, and one week after the procedure. We hypothesize that there will be no significant difference in pain levels between the two treatment approaches. The results will help dentists decide the best treatment plan for their diabetic patients without worrying about causing more pain.

ELIGIBILITY:
Inclusion Criteria:Patients aged between 12 and 60 years.

Diagnosed with Type 1 or Type 2 Diabetes Mellitus.

In need of root canal treatment on a single-rooted tooth.

A clinical diagnosis of either irreversible pulpitis or necrotic pulp in the indicated tooth.

Willingness and ability to understand and provide written informed consent (and assent with parental consent for minors).

-

Exclusion Criteria:

* Pregnancy.

Known history of allergy to local anesthetics.

Presence of large periapical radiolucent lesions (typically defined as >5mm in diameter).

Current use of long-term analgesic or anti-inflammatory medication (which could alter pain perception).

Teeth with complex root canal anatomy (e.g., calcified canals, C-shaped canals) that would complicate standard treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Moderate-to-Severe Pain at 24 Hours Post-Operation | 24 Hours after the procedure
  Measurement Tool: Numeric Rating Scale (NRS), an 11-point scale from 0 (no pain) to 10 (worst imaginable pain).
  Unit of Measure: Percentage (%) of patients.
  Description: The proportion of patients reporting a pain intensity score of 4 or greater on the NRS during movement (e.g., coughing or ambulation) at the 24-hour post-operative time point.

SECONDARY OUTCOMES:
Mean Resting Pain Intensity at 24 Hours Post-Operation | 24 hours after the procedure
  Measurement Tool: Numeric Rating Scale (NRS), an 11-point scale from 0 (no pain) to 10 (worst imaginable pain).
  Unit of Measure: Percentage (%) of patients.
  Description: The proportion of patients reporting a pain intensity score of 4 or greater on the NRS during movement (e.g., coughing or ambulation) at the 24-hour post-operative time point.

IPD SHARING:
Plan to Share IPD: No